CLINICAL TRIAL: NCT04488913
Title: Rapid Acute Coronary Syndrome Exclusion Using the Beckman Coulter Access High-sensitivity I Troponin
Brief Title: Rapid Acute Coronary Syndrome Exclusion Using High-sensitivity I Troponin
Acronym: RACE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Beckman Coulter, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Miller, MD, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: pending
Record Dates: First submitted 2020-07-19; First posted 2020-07-28 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Chest Pain; Myocardial Ischemia
Keywords: high-sensitivity troponin; chest pain
MeSH Terms: conditions — Chest Pain; Myocardial Ischemia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge Cluster Randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Treatment (Other): Exposure to traditional evaluation for suspected acute coronary syndrome (ACS) with ECG, 0- and 3-hour troponin testing using the 99th percentile as the upper reference limit, and application of the History, EKG, Age, Risk factors, and troponin (HEART) score.
  Interventions: Other: Standard of Care
- RACE-IT pathway (Active Comparator): Exposure to new protocol for suspected ACS, which includes the use of 0- and 1-hour ECG and high-sensitivity troponin testing and application of the HEAR score (a modification of the HEART score)
  Interventions: Other: RACE-IT Pathway

INTERVENTIONS:
Other: RACE-IT Pathway — This care pathway includes the evaluation of suspected acute coronary syndrome with high-sensitivity troponin I testing and further prognostication as needed with a modified HEART score
  Arms: RACE-IT pathway
Other: Standard of Care — Standard of care protocol that uses the 99th percentile troponin values for evaluation of suspected acute coronary syndrome and further prognostication using the HEART score
  Arms: Standard of Care Treatment

SUMMARY:
As part of the planned implementation of a new clinical pathway using hs-cTnI, the investigators will measure patient outcomes and clinical processes in a real-world scenario throughout an integrated health system across 9 emergency departments (ED).

DETAILED DESCRIPTION:
This is a pragmatic, implementation study testing the implications of a real-world execution of a rapid evaluation pathway for suspected ACS using the Beckman hs-cTnI assay. As the new protocol is executed across 9 EDs within an integrated health system, the investigators will study its effects on patient and system-level metrics. A modified stepped wedge design will be utilized that allows comparison of the RACE-IT pathway with standard of care management

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old presenting to the ED for whom a treating clinician suspects ACS and orders a baseline ECG and cardiac troponin.

Exclusion Criteria:

1. ST-segment Myocardial Infarction (STEMI) leading to immediate reperfusion therapy
2. Any ED-drawn hs-cTnI value > 99th percentile (18 ng/L)
3. Clear traumatic cause for symptoms (e.g., direct chest wall trauma, motor vehicle accident)
4. A transfer from another facility
5. Primary residence outside the state of Michigan
6. Previous inclusion in the study
7. Enrolled in hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32609 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Safe ED discharge | 30 days after initial presentation
  Proportion of patients with safe discharges home from the ED, defined as being without death or acute myocardial infarction within 30-days

SECONDARY OUTCOMES:
Length of hospital stay | From date and time of start of emergency department encounter until date and time of end of ED or hospital encounter (whichever is latest), assessed up to 7 days.
  Length of time from initial presentation to the Emergency Department until final discharge from the Emergency Department or Observation Unit
Number of participants with death or acute myocardial infarction | 30-day and through 1 year
  Death or presence of acute myocardial infarction determined by adjudication panel
Number of participants with revascularization or rehospitalization for cardiovascular disease | 30-days
  revascularization includes percutaneous coronary interventions and rehospitalization is inclusive of any such event for acute heart failure, acute myocardial infarction, or arrhythmia
Composite number of cardiology resources utilized | 30-days
  Cardiology resources are inclusive of completed orders for cardiac stress tests, cardiology consultation, coronary computed tomography, coronary angiography, and percutaneous coronary intervention
Hospital payments received | 30-days
  The total hospital payments received for the initial ED visit and any subsequent hospitalizations and procedures that are cardiology related over 30-days from the initial encounter.

OTHER OUTCOMES:
Pre-specified sub-group analyses of the primary outcome | 30 days
  We will explore analysis assessing gender-specific cut-points for hs-cTnI associated with safe discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Derived] Miller J, Cook B, Gunaga S, Fadel R, Gandolfo C, Emakhu J, Mills NL, Mahler S, Levy P, Parikh S, Krupp S, Hawatian K, Nour K, Klausner H, Gindi R, Hudson M, Perrotta G, Zweig B, Lanfear D, Kim H, Danagoulian S, Keerie C, Nassereddine H, Morton T, Affas Z, Husain A, McCord J; RACE-IT Research Group. Health Care Resource Utilization for Patients With Suspected Myocardial Infarction: A Secondary Analysis of the RACE-IT Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e256930. doi: 10.1001/jamanetworkopen.2025.6930. PMID 40279128
- [Derived] Glintborg D, Moller JK, Rubin KH, Lidegaard O, T'Sjoen G, Larsen MJO, Hilden M, Lehmann Christensen L, Andersen MS. Mental and Physical Health Among Danish Transgender Persons Compared With Cisgender Persons. JAMA Netw Open. 2025 Apr 1;8(4):e257115. doi: 10.1001/jamanetworkopen.2025.7115. PMID 40272800
- [Derived] Miller J, Cook B, Singh-Kucukarslan G, Tang A, Danagoulian S, Heath G, Khalifa Z, Levy P, Mahler SA, Mills N, McCord J. RACE-IT - Rapid Acute Coronary Syndrome Exclusion using the Beckman Coulter Access high-sensitivity cardiac troponin I: A stepped-wedge cluster randomized trial. Contemp Clin Trials Commun. 2021 Apr 23;22:100773. doi: 10.1016/j.conctc.2021.100773. eCollection 2021 Jun. PMID 34013092